#### **Analysis Plan for the NORA Study**

#### **Introduction:**

This analysis plan integrates analyses suggested by the investigators as well as requests by regulatory authorities and the independent Safety Monitoring and Advisory Council (SMAC).

The primary objective of this one-arm, non-comparative study is to investigate the frequency of insertion-, localization and removal-related events.

In principle, three different sets of analyses could be provided:

- 1) the 'as treated' (AT) population and
- 2) the 'intention to treat' (ITT) population
- 3) the 'per protocol' population

However, in this one-arm study AT and ITT populations will be almost identical. A woman who is included in the study will only be exposed to one treatment (Nexplanon). Therefore, the true exposure (AT) will be identical with the intended exposure (ITT). The only theoretical exception would be a woman where no insertion attempt is made although the woman agreed to participate. The inclusion of those women into the ITT analysis set would dilute the rate of insertion- and removal-related adverse events. I.e., the ITT analysis would slightly underestimate the risk associated with the use of Nexplanon. Therefore, an ITT analysis will not be done.

Also 'per protocol' analyses will not be done, because 1) there are no medical inclusion and exclusion criteria in this non-interventional study, and 2) protocol violations against non-medical inclusion and/or exclusion criteria (such as enrollment of a woman who refuses to sign the informed consent form) will lead to immediate exclusion of the participant. Therefore, the results of the 'per protocol' analysis would be identical with the AT analysis.

It is conceivable that women, who had a previous implant (repeat / consecutive users previously using Implanon or Norplant) might differ in their reporting of adverse events and might be at lower risk for insertion, localization and or removal associated events from women who never used a hormonal implant before (first-time users). Therefore, the analyses will include three analysis subsets:

- 1) all users
- 2) first-time users ("starter")
- 3) repeat/consecutive users

<u>Section A</u> of this statistical analysis plan will provide a description of the population (total study population and stratified by first time users and repeat/consecutive users) and the availability of follow-up information. Three of the tables in this section (Tables A3a, A3b, A4) have the HCP as unit, not the woman.

<u>Section B</u> shows descriptive tables of baseline characteristics and potential prognostic factors in the different user cohort

<u>Section C</u> shows descriptive tables of the outcomes of interest. Characterization of the frequency of specific insertion-, localization- and removal-related events among Nexplanon users under standard clinical practice will mostly be undertaken via point-estimates of the event rate as well as 95% confidence intervals. The impact of potential prognostic factors will be analyzed using multivariate regression models and/or stratified analyses.

Potential prognostic factors for the outcomes of interest include e.g. age (< 30 y vs. ≥30), BMI (<30 vs. ≥30), user status (first time users vs. repeat users), experience of healthcare professional with Implanon insertions in the past year (<10/y vs. >=10/y) and Nexplanon insertions in total (<5 NXPL vs. >=5 NXPL). The cut-off point regarding experience of the healthcare professional were chosen arbitrary, sensitivity analyses with different cut-off points will done. Additional prognostic factors and classification categories might be added on request of regulatory authorities or the Safety Monitoring and Advisory Board.

This statistical analysis plan will be the basis for the final analysis of the data at study end.

The bi-annual interim report will show data reflected in the tables A1, A3-4, B1-13, C1, C3-11, depending on the status of the study – no data on localization / removal and post-removal questions are expected during the first year of the study.

At study end all tables in the B section will be used to compare characteristics of women who remain during follow-up vs. those who are who dropped out before removal or were Lost to Follow-up.

In case of Loss to FU and drop out before removal exposure to Nexplanon will be based on the last available FU information.

Number of missing answers will be presented in the tables but percentages and confidence intervals will be based on the total number of non-missing answers.

#### List of abbreviations

AT As Treated

BMI Body Mass Index

CI Confidence Interval

FU Follow-up

HC Hormonal Contraceptive

HCP Health Care Professional

ITT Intention to Treat

L/R Localization / Removal

Miss Missing

n Number

NXPL Nexplanon

OC Oral Contraceptive

Pl Pearl Index (pregnancies per 100 WY)

RR Relative Risk

(S)AE (Serious) Adverse Event

WY Women Years (one WY = 365.25 days of exposure)

### Section A: Number of study participants, User Status and Follow-up

#### Table A1. Number of women included in the study (Date of analysis: . . .)

Table A1-1 - Women included in the study by user Type, Complete Cohort

| | n | % |
|--------------------------|---|---|
| First time users | | |
| Repeat/Consecutive users | | |
| Total number at baseline | | |

#### Table A2. Drop-outs and loss to follow-up (Date of analysis: . . .)

Table A2-1 Complete Cohort

| | | | Follow-up | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | Baseline | FU1 | FU2 | FU3 | FU4 | FU5 | Localization<br>/ Removal<br>FU | Post<br>removal<br>FU | Total |
| No of women with available information per period | | | | | | | | | |
| No of women who got their Implant removed (%) | | | | | | | | | |
| No of drop outs (%) | | | | | | | | | |
| No. of women who are lost to follow-up (%) | | | | | | | | | |

Table A2-2 First time users only (format see Table A2-1)

Table A2-3 Repeat/Consecutive users only (format see Table A2-1)

Table A3. Number healthcare professionals by categories of experience in Implanon/Nexplanon insertions (Date of analysis: . . .)

Table A3 a Implant insertions in the past year

| Implanon insertions in the past year | N | % |
|--------------------------------------|---|---|
| <5 in the past year | | |
| >=5 - <10 in the past year | | |
| >= 10 in the past year | | |
| Miss <sup>#</sup> | | |
| Total | | |

Table A3 b Total number of Nexplanon insertions

| Total number of Nexplanon insertions | N | % |
|--------------------------------------|---|---|
| <5 | | |
| >=5 - <10 | | |
| >= 10 | | |
| Miss# | | |
| Total | | |

# number of missing answers are presented, percentages based only on the total number of non-missing answers

 Table A4.
 Educational background of Healthcare Professional (Date of analysis: . . .)

| | N | % |
|--------------------|---|---|
| Nurse | | |
| Nurse Practitioner | | |
| Gynecologist | | |
| Other* | | |
| Miss <sup>#</sup> | | |
| Total | | |

<sup>\*</sup>If another educational background of HCP shown in the "Other" category accounts for more then 1% of the Nexplanon insertions in the study, it will be listed in a separate category

<sup>#</sup> number of missing answers are presented, percentages based only on the total number of non-missing answers

### **Section B: Demographics**

#### Table B1. Age (y), weight (lb) and BMI at study entry (Date of analysis: . . .)

Table B1-1 Complete Cohort

| | NXPL |
|-----------------------|------|
| Age, Mean [SD] | |
| Age, Minimum | |
| Age, Percentile 5 | |
| Age, Percentile 25 | |
| Age, Median | |
| Age, Percentile 75 | |
| Age, Percentile 95 | |
| Age, Maximum | |
| Weight, Mean [SD] | |
| Weight, Minimum | |
| Weight, Percentile 5 | |
| Weight, Percentile 25 | |
| Weight, Median | |
| Weight, Percentile 75 | |
| Weight, Percentile 95 | |
| Weight, Maximum | |
| Weight, Miss | |
| BMI, Mean [SD] | |
| BMI, Minimum | |
| BMI, Percentile 5 | |
| BMI, Percentile 25 | |
| BMI, Median | |
| BMI, Percentile 75 | |
| BMI, Percentile 95 | |
| BMI, Maximum | |
| BMI, Miss | |

Table B1-2 First time users only (format see Table B1-1)
Table B1-3 Repeat/Consecutive users only (format see Table B1-1)

 Table B2.
 Age and BMI distribution (Date of analysis: . . .)

Table B2-1 Complete Cohort

| | n | % | 95% CI |
|-------------------|---|---|--------|
| Age category | | | |
| <20 | | | |
| 20-29 | | | |
| 30-39 | | | |
| 40-49 | | | |
| >=50 | | | |
| TOTAL | | | |
| BMI category | | | |
| BMI <20 | | | |
| BMI >=20 & <25 | | | |
| BMI >=25 & <30 | | | |
| BMI >=30 & <35 | | | |
| BMI >=35 | | | |
| Miss# | | | |
| TOTAL | | | |
| Weight category | | | |
| <88 lb | | | |
| 88-<110 lb | | | |
| 110-<132 lb | | | |
| 132-<154 lb | | | |
| 154-<176 lb | | | |
| 176-<198 lb | | | |
| 198-<220 lb | | | |
| >= 220 lb | | | |
| Miss <sup>#</sup> | | | |
| TOTAL | | | |

<sup>#</sup> number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

Table B2-2 First time users only (format see Table B2-1)

Table B2-3 Repeat/Consecutive users only (format see Table B2-1)

Table B3. Proportion of Women who have ever been pregnant, had a delivery in the last 12 months, and who had Miscarriage / Abortion in the last 12 months (Date of analysis: . . .)

Table B3-1 Complete Cohort

| | n | % | 95% CI |
|--------------------------------------------------|---|---|--------|
| Ever pregnant | | | |
| Yes | | | |
| No | | | |
| Miss* | | | |
| Delivery within the last 12 months | | | |
| Yes | | | |
| No | | | |
| Miss <sup>#</sup> | | | |
| Miscarriage / Abortion within the last 12 months | | | |
| Yes | | | |
| Of which | | | |
| First trimester miscarriage / abortion | | | |
| Second trimester miscarriage / abortion | | | |
| No | | | |
| Miss <sup>#</sup> | | | |

<sup>#</sup> number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

Table B3-2 First time users only (format see Table B3-1)

Table B3-3 Repeat/Consecutive users only (format see Table B3-1)

#### Table B4. Age at menarche, number of live births (Date of analysis: . . .)

#### Table B4-1 Complete Cohort

| | NXPL |
|--------------------------------------|------|
| Age at Menarche, Mean [SD] | |
| Age at Menarche, Minimum | |
| Age at Menarche, Percentile 5 | |
| Age at Menarche, Percentile 25 | |
| Age at Menarche, Median | |
| Age at Menarche, Percentile 75 | |
| Age at Menarche, Percentile 95 | |
| Age at Menarche, Maximum | |
| Age at Menarche, Miss | |
| Number of Live Births, Mean [SD] | |
| Number of Live Births, Minimum | |
| Number of Live Births, Percentile 5 | |
| Number of Live Births, Percentile 25 | |
| Number of Live Births, Median | |
| Number of Live Births, Percentile 75 | |
| Number of Live Births, Percentile 95 | |
| Number of Live Births, Maximum | |
| Number of Live Births, Miss | |

Table B4-2 First time users only (format see Table B4-1)

Table B4-3 Repeat/Consecutive users only (format see Table B4-1)

#### Table B5. Implant History (Date of analysis: . . .)

Table B5-1 Complete Cohort

| | n | % | 95% CI |
|-----------------------------------------------|---|---|--------|
| Ever contraceptive Implant before study entry | | | |
| Yes | | | |
| No | | | |
| Miss* | | | |
| Total duration of Implant use | | | |
| <=1 year | | | |
| >1 & <=5 years | | | |
| >5 & <=10 years | | | |
| >10 years | | | |
| Miss | | | |

# number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

#### Table B6. Hormonal Contraception History (Date of analysis: . . .)

Table B6-1 Complete Cohort

| | n | % | 95% CI |
|------------------------------------------|---|---|--------|
| Ever OC / HC Use | | | |
| Yes | | | |
| No | | | |
| Miss# | | | |
| Number of months since last OC / HC use§ | | | |
| <=3 months ago | | | |
| >3 & <=6 months ago | | | |
| >6 & <=12 months ago | | | |
| >12 months ago | | | |
| Miss# | | | |
| Total duration of OC / HC use | | | |
| <=1 year | | | |
| >1 & <=5 years | | | |
| >5 & <=10 years | | | |
| >10 years | | | |
| Miss* | | | |

<sup>#</sup> number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

Table B6-2 First time users only (format see Table B6-1)

Table B6-3 Repeat/Consecutive users only (format see Table B6-1)

<sup>§</sup> For hormonal injections the day the next injection would have been due is used for determination of number of months since last HC use

#### Table B7. Smoking Status (Date of analysis: . . .)

Table B7-1 Complete Cohort

| | n | % | 95% CI |
|---------------------------------------|---|---|--------|
| Never smoker | | | |
| Current smoker | | | |
| Thereof | | | |
| Heavy Smoker (>15 cigarettes per day) | | | |
| Ex-Smoker | | | |
| Thereof | | | |
| Heavy Smoker (>15 cigarettes per day) | | | |
| Miss# | | | |

# number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

Table B7-2 First time users only (format see Table B7-1)

Table B7-3 Repeat/Consecutive users only (format see Table B7-1)

#### Table B8. Number of Cigarettes (Date of analysis: . . .)

Table B8-1 Complete Cohort

| | Current<br>Smoker | Ex-Smoker |
|-------------------------------------|-------------------|-----------|
| Number of Cigarettes, Mean [SD] | | |
| Number of Cigarettes, Minimum | | |
| Number of Cigarettes, Percentile 5 | | |
| Number of Cigarettes, Percentile 25 | | |
| Number of Cigarettes, Median | | |
| Number of Cigarettes, Percentile 75 | | |
| Number of Cigarettes, Percentile 95 | | |
| Number of Cigarettes, Maximum | | |
| Number of Cigarettes, Miss | | |

Table B8-2 First time users only (format see Table B8-1)

Table B8-3 Repeat/Consecutive users only (format see Table B8-1)

#### Table B9. Educational Level (Date of analysis: . . .)

Table B9-1 Complete Cohort

| | n | % | 95%<br>CI |
|----------------------------------------------------|---|---|-----------|
| Elementary School (at most 5 year) | | | |
| Junior High or Middle School (at most 8 years) | | | |
| High school (at most 12 years) | | | |
| Some college/Associate's Degree/Technical training | | | |
| College/University Bachelor Degree | | | |
| Post-College/University or higher | | | |
| Miss# | | | |

<sup>#</sup> number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

Table B9-2 First time users only (format see Table B9-1)

Table B9-3 Repeat/Consecutive users only (format see Table B9-1)

## Table B10. Self-reported history of selected diseases at baseline: Absolute numbers of reports and crude prevalence (%) (Date of analysis: ...)

Table B10-1 Complete Cohort

| | n | % | 95%<br>CI |
|------------------------------------|---|---|-----------|
| Medical History | | | |
| Venous thromboembolism (DVT or PE) | | | |
| Myocardial Infarction | | | |
| Stroke | | | |
| Cancer* | | | |
| Other serious diseases | | | |
| Operations | | | |

<sup>\*</sup> sub-category will be shown for cancer types with more than 5 reports

Table B10-2 First time users only (format see Table B10-1)

Table B10-3 Repeat/Consecutive users only (format see Table B10-1)

#### Table B11 Use of local anesthetic and insertion site (Date of analysis: . . .)

Table B11-1 Complete Cohort

| | n | % | 95%<br>CI |
|----------------------------------------------|---|---|-----------|
| Local Anesthetic | | | |
| Yes | | | |
| No | | | |
| Miss# | | | |
| Implant inserted in the non-<br>dominant arm | | | |
| Yes | | | |
| No | | | |
| Miss <sup>#</sup> | | | |
| Position of implant | | | |
| Over biceps muscle | | | |
| Over triceps muscle | | | |
| In sulcus bicipitalis medialis | | | |
| Other | | | |
| Miss# | | | |

<sup>#</sup> number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

#### Additional categories may be added for exploratory reasons

Table B11-2 First time users only (format see Table B11-1)

Table B11-3 Repeat/Consecutive users only (format see Table B11-1)

### Section C: Outcomes of interest

#### Table C1. Duration of Nexplanon use in Years (Date of analysis: . . .)

Table C1-1 Complete Cohort

| | NXPL |
|--------------------------------|------|
| Duration of use, Mean [SD] | |
| Duration of use, Minimum | |
| Duration of use, Percentile 5 | |
| Duration of use, Percentile 25 | |
| Duration of use, Median | |
| Duration of use, Percentile 75 | |
| Duration of use, Percentile 95 | |
| Duration of use, Maximum | |
| Duration of use, Miss | |

Table C1-2 First time users only (format see Table C1-1)

Table C1-3 Repeat/Consecutive users only (format see Table C1-1)

#### Table C2. Implant palpability reported by the woman (Date of analysis: ...)

Table C2-1 Complete Cohort

| | | | Follow-up | | | | |
|---|---|---|---|---|---|---|---|
| | Insertion | FU1 | FU2 | FU3 | FU4 | FU5 | Localization /<br>Removal FU* |
| Women who could feel implant (%) | | | | | | | |
| Women who could not feel implant (%) | | | | | | | |
| Missing information (%) | | | | | | | |

<sup>\*</sup> reported by HCP

Table C2-2 First time users only (format see Table C2-1)

Table C2-3 Repeat/Consecutive users only (format see Table C2-1)

Table C2-4 BMI <20 (format see Table C2-1)

Table C2-5 BMI >=20 - <30 (format see Table 2-1)

Table C2-6BMI >=30 (format see Table C2-1)

**Table C3.** Validated¹ insertion related complications reported by the woman: Absolute numbers of reports and incidence proportion (per 1,000 insertions) (Date of analysis: . . .)

Table C3-1 Complete Cohort

| C3-1 Complete Conort | | Incidence | / |
|---|---|---|---|
| | n | Proportion* | 95% CI |
| Severe Pain | | | |
| reported: | | | |
| At Baseline | | | |
| At FU | | | |
| At / After Removal | | | |
| Injury to blood vessels or blood clots in the arm | | | |
| reported: | | | |
| At Baseline | | | |
| At FU | | | |
| At / After Removal | | | |
| Pins and needles /<br>numbness in the arm /<br>hand / fingers | | | |
| reported: | | | |
| At Baseline | | | |
| At FU | | | |
| At / After Removal | | | |
| Altered strength / movement in the arm | | | |
| reported: | | | |
| At Baseline | | | |
| At FU | | | |
| At / After Removal | | | |

<sup>\*</sup> per 1,000 insertions

<sup>&</sup>lt;sup>1</sup> Validated means that for a self-reported event / complaint by the women further information is collected from the woman and the treating physician or hospital to confirm the validity of the information

#### Additional categories may be added for complications

Table C3-2 First time users only (format see Table C3-1)

Table C3-3 Repeat/Consecutive users only (format see Table C3-1)

Table C3-4 BMI <20 (format see Table C3-1)

Table C3-5 BMI  $\geq$  20 -  $\leq$  30 (format see Table 3-1)

Table C3-6 BMI >=30 (format see Table C3-1)

Table C3-7 Age <30 (format see Table C3-1)

Table C3-8 Age >=30 (format see Table C3-1)

Table C3-9 Experience of Physician <10 Implanon insertions in the past year (format see Table C3-1)

Table C3-10 Experience of Physician >=10 Implanon insertions in the past year (format see Table C3-1)

Table C3-11 Experience of Physician <5 Nexplanon insertions in total (format see Table C3-1)

Table C3-12 Experience of Physician >= 5 Nexplanon insertions in total (format see Table C3-1)

# Table C4. Any significant issues during insertion procedure insertion / insertion attempt (reported by HCP): absolute number and incidence proportion (per 1.000 insertions) (Date of analysis: . . .)

Table C4-1 Complete Cohort

| Category | n | Incidence<br>Proportion* | 95%CI |
|---|---|---|---|
| Insertion successful | | | |
| Yes, first attempt successful | | | |
| Yes, but multiple insertion attempts required (i.e. at least 1 unsuccessful insertion) | | | |
| No, implant insertion unsuccessful | | | |
| Any significant issues during insertion procedure of which | | | |
| Difficulty removing protection cap | | | |
| Difficulty sliding needle to its full length into skin | | | |
| Needle stick injury | | | |
| Difficulty unlocking purple slider | | | |
| Needle inserted too deep | | | |
| Difficulty moving purple slider fully to the back | | | |
| Needle inserted too superficial | | | |
| Implant (partially) sticks out of skin after insertion | | | |
| Injury to nerve or blood-vessel | | | |
| Needle visible after insertion (not fully retracted) | | | |
| Other | | | |
| Miss | | | |

<sup>\*</sup> per 1,000 insertions

#### Additional categories may be added for complications

Table C4-2 First time users only (format see Table C4-1)
Table C4-3 Repeat/Consecutive users only (format see Table C4-1)

Table C4-4 BMI <20 (format see Table C4-1)

```
Table C4-5 BMI >=20 - <30 (format see Table 4-1)
Table C4-6 BMI >=30 (format see Table C4-1)
```

Table C4-7 Age <30 (format see Table C4-1)

Table C4-8 Age >=30 (format see Table C4-1)

Table C4-9 Experience of Physician <10 Implanon insertions in the past year (format see Table C4-1)

Table C4-10 Experience of Physician >=10 Implanon insertions in the past year (format see Table C4-1)

Table C4-11 Experience of Physician <5 Nexplanon insertions in total (format see Table C4-1) Table C4-12 Experience of Physician >=5 Nexplanon insertions in total (format see Table C4-1)

# Table C5. Localization procedures (reported by HCP): Absolute numbers of reports and incidence proportion (per 1,000 insertions) (Date of analysis: . . .)

Table C5-1 Complete Cohort

| | n | Incidence<br>Proportion* | 95% CI |
|----------------------------|---|--------------------------|--------|
| Implant not palpable | | | |
| reported: | | | |
| At Insertion | | | |
| At L/R | | | |
| Any Localization procedure | | | |
| No | | | |
| Yes | | | |
| If Yes, reported: | | | |
| At Insertion | | | |
| At L/R | | | |
| X-Ray | | | |
| reported: | | | |
| At Insertion | | | |
| At L/R | | | |
| Ultrasound | | | |
| reported: | | | |
| At Insertion | | | |
| At L/R | | | |
| СТ | | | |
| reported: | | | |
| At Insertion | | | |
| At L/R | | | |
| MRI | | | |
| reported: | | | |
| At Insertion | | | |
| At L/R | | | |

Table C5-1 continued

| C5-1 continued | ı <b>ı</b> | ! | i 1 |
|---|---|---|---|
| Hormone Assay (ENG) | | | |
| reported: | | | |
| At Insertion | | | |
| At L/R | | | |
| ENG detected | | | |
| ENG not detected | | | |
| ENG Result pending | | | |
| Implant migration (at L/R) | | | |
| Yes | | | |
| No | | | |
| Location of Implant (at Insertion) | | | |
| Dermal | | | |
| Subdermal connective | | | |
| tissue | | | |
| Adjacent to the fascial tissue | | | |
| Within the muscle | | | |
| Not determined | | | |
| Miss | | | |
| Location of Implant (at L/R) | | | |
| Dermal | | | |
| Subdermal connective | | | |
| tissue | | | |
| Adjacent to the fascial tissue | | | |
| Within the muscle | | | |
| Not determined | | | |
| Miss | | | |
| Hospitalization needed for localization procedure (L/R) | | | |
| Yes | | | |
| No | | | |
| 1 | | | ! I |

#### Table C5-1 continued



\*per 1,000 insertions

A woman can have more than one localization procedure during the study period, and also the same localization procedure more than one time

#### Additional categories may be added

```
Table C5-2 First time users only (format see Table C5-1)
```

Table C5-3 Repeat/Consecutive users only (format see Table C5-1)

Table C5-4 BMI <20 (format see Table C5-1)

Table C5-5 BMI >=20 - <30 (format see Table 5-1)

Table C5-6 BMI >=30 (format see Table C5-1)

Table C5-7 Age <30 (format see Table C5-1)

Table C5-8 Age >=30 (format see Table C5-1)

Table C5-9 Experience of Physician <10 Implanon insertions in the past year (format see Table C5-1)

Table C5-10 Experience of Physician >=10 Implanon insertions in the past year (format see Table C5-1)

Table C5-11 Experience of Physician <5 Nexplanon insertions in total (format see Table C5-1)

Table C5-12 Experience of Physician >= 5 Nexplanon insertions in total (format see Table C5-1)

### Table C6. Number of Women with non-palpable Implant and related Localization Procedures (Date of analysis: . . .)

Table C6-1 Complete Cohort

| | n | % | 95% CI |
|-----------------------------|---|---|--------|
| Implant inserted | | | |
| thereof | | | |
| Implant not palpable by HCP | | | |
| thereof | | | |
| Any Localization procedure | | | |
| thereof | | | |
| X-Ray | | | |
| Thereof Implant localized | | | |
| Ultrasound | | | |
| Thereof implant localized | | | |
| СТ | | | |
| Thereof implant localized | | | |
| MRI | | | |
| Thereof implant localized | | | |
| Hormone Assay (ENG) | | | |
| Thereof ENG positive | | | |

```
Table C6-2 First time users only (format see Table C6-1)
Table C6-3 Repeat/Consecutive users only (format see Table C6-1)
```

Table C6-4 BMI <20 (format see Table C6-1)

Table C6-5 BMI >=20 - <30 (format see Table C6-1)

Table C6-6 BMI >=30 (format see Table C6-1)

Table C6-7 Age <30 (format see Table C6-1)

Table C6-8 Age >=30 (format see Table C6-1)

Table C6-9 Experience of Physician <10 Implanon insertions in the past year (format see Table C6-1)

Table C6-10 Experience of Physician >=10 Implanon insertions in the past year (format see Table C6-1)

Table C6-11 Experience of Physician <5 Nexplanon insertions in total (format see Table C6-1) Table C6-12 Experience of Physician >=5 Nexplanon insertions in total (format see Table C6-1)

## Table C7. Complications during removal: Absolute numbers of reports and Incidence Proportion (per 1,000 insertions) (Date of analysis: ...)

Table C7-1 Complete Cohort

| | | n | Prop* | 95% CI |
|---|---|---|---|---|
| Implant removed | | | | |
| | Yes | | | |
| | No | | | |
| Any Complications during removal (attempt) | | | | |
| | No | | | |
| | Yes | | | |
| thereof | | | | |
| Injury to nerve/blood vessel | | | | |
| Implant located near nerve and/or blood vessel | | | | |
| Implant encased in fibrotic tissue making removal difficult | | | | |
| Implant located too deep | | | | |
| Implant migrated | | | | |
| Implant not found | | | | |
| Multiple attempts required | | | | |
| Others | | | | |
| Additional surgical procedure required | | | | |
| | Yes | | | |
| | No | | | |
| Local anesthesia used | | | | |
| General anesthesia used | | | | |
| Ocheral and stricts a decu | | | | |
| Hospitalization for removal | | | | |
| | Yes | | | |
| | No | | | |
| *per 1.000 insertions | | 1 | | |

\*per 1,000 insertions

#### Additional categories may be added for complications

Table C7-2 First time users only (format see Table C7-1)

Table C7-3 Repeat/Consecutive users only (format see Table C7-1)

Table C7-4 BMI <20 (format see Table C7-1)

Table C7-5 BMI  $\geq$  20 -  $\leq$  30 (format see Table C7-1)

Table C7-6 BMI >=30 (format see Table C7-1)

Table C7-7 Age <30 (format see Table C7-1)

Table C7-8 Age >=30 (format see Table C7-1)

Table C7-9 Experience of Physician <10 Implanon insertions in the past year (format see Table C7-1)

Table C7-10 Experience of Physician >=10 Implanon insertions in the past year (format see Table C7-1)

Table C7-11 Experience of Physician <5 Nexplanon insertions in total (format see Table C7-1)

Table C6-12 Experience of Physician >= 5 Nexplanon insertions in total (format see Table C7-1)

### Table C8: Pregnancies: Absolute numbers of reports and Pearl Index (per 100 WY) (Date of analysis: . . .)

Table C8-1 Complete Cohort

| Category | n | PI* | 95%CI |
|---|---|---|---|
| Total Pregnancies | | | |
| thereof | | | |
| Pre-Treatment Pregnancies | | | |
| In-Treatment Pregnancies | | | |
| thereof | | | |
| Taking concurrent medication with potential interaction | | | |
| Post-Treatment Pregnancies <sup>2</sup> | | | |
| Thereof | | | |
| With an estimated date of conception 1-7 days after removal | | | |
| With an estimated date of conception 8-14 days after removal | | | |
| With an estimated date of conception more than 14 days after removal | | | |
| Non-insertion Pregnancies | | | |

<sup>\*</sup> pregnancies per 100 WYs of exposure3

Table C8-2 First time users only (format see Table C8-1)

Table C8-3 Repeat/Consecutive users only (format see Table C8-1)

Table C8-4 BMI <20 (format see Table C8-1)

Table C8-5 BMI  $\geq$  20 -  $\leq$  30 (format see Table C8-1)

Table C8-6 BMI >=30 (format see Table C8-1)

Table C8-7 Body weight <155lb only (format see Table C8-1)

Table C8-8 Body weight >=155lb only (format see Table C8-1)

Table C8-9 Age <30 only (format see Table C8-1)

Table C8-10 Age >=30 only (format see Table C8-1)

<sup>&</sup>lt;sup>2</sup> For Post-Treatment Pregnancies the PI calculation does always include the In-treatment pregnancies and (if applicable) pregnancies from the previous Post-treatment Period

<sup>&</sup>lt;sup>3</sup> Nexplanon exposure: time from insertion day to estimated conception day or, in case of post-removal pregnancies, the day of Nexplanon removal

#### Table C9: Outcomes of Pre-, In- and Post-Treatment Pregnancies (Date of analysis: ...)

Table C9-1 Complete Cohort

| Category | n | % | 95%CI |
|---|---|---|---|
| Outcome of Pre-Treatment Pregnancy | | | |
| Healthy child | | | |
| Induced abortion | | | |
| Spontaneous abortion | | | |
| Ectopic Pregnancy | | | |
| Malformation | | | |
| Outcome of In-Treatment Pregnancy | | | |
| Healthy child | | | |
| Induced abortion | | | |
| Spontaneous abortion | | | |
| Ectopic Pregnancy | | | |
| Malformation | | | |
| Outcome of Post-Treatment Pregnancy | | | |
| With an estimated date of conception1-7 days after removal | | | |
| Healthy child | | | |
| Induced abortion | | | |
| Spontaneous abortion | | | |
| Ectopic Pregnancy | | | |
| Malformation | | | |
| With an estimated date of conception<br>8-14 days after removal | | | |
| Healthy child | | | |
| Induced abortion | | | |
| Spontaneous abortion | | | |
| Ectopic Pregnancy | | | |
| Malformation | | | |
| Malformation | | | |

```
Table C9-2 First time users only (format see Table C9-1)
Table C9-3 Repeat/Consecutive users only (format see Table C9-1)
```

Table C9-4 BMI <20 (format see Table C9-1)

Table C9-5 BMI >=20 - <30 (format see Table C9-1)

Table C9-6 BMI >=30 (format see Table C9-1)

Table C9-7 Body weight <155lb only (format see Table C9-1)
Table C9-8 Body weight >=155lb only (format see Table C9-1)

Table C9-9 Age <30 only (format see Table C9-1)
Table C9-10 Age >=30 only (format see Table C9-1)

#### Table C10-Reasons for removing the Implant (Date of analysis: ...)

Table C10-1 Complete Cohort

| Event category | n | % | 95% CI |
|----------------------------------------------------------|---|---|--------|
| The implant had been in place for at least 3 years | | | |
| Planning pregnancy and/or contraception no longer needed | | | |
| Became pregnant despite Nexplanon use | | | |
| Problem with implant | | | |
| Menstrual/bleeding problems | | | |
| Miss <sup>#</sup> | | | |

<sup>#</sup> number of missing answers are presented, percentages and confidence intervals based only on the total number of non-missing answers

#### Additional categories may be added for reasons

Table **C10**-2 First time users only (format see Table **C10**-1)
Table **C10**-3 Repeat/Consecutive users only (format see Table **C10**-1)

Table **C10**-4 BMI <20 (format see Table **C10**-1)

Table **C10**-5 BMI >=20 - <30 (format see Table **C10**-1)

Table **C10**-6 BMI >=30 (format see Table **C10**-1)

Table C10-7 Age <30 (format see Table C10-1)

Table C10-8 Age >=30 (format see Table C10-1)

# Table C11- Validated SAEs not related to insertion-, localization- or removal-procedure of Nexplanon: Absolute numbers of reports and incidence rate (per 10,000 WY of exposure) (Date of analysis: ...)

#### Table C11-1 Complete Cohort

| Event category | n | Incidence<br>Rate* | 95% CI |
|--------------------------|---|--------------------|--------|
| Cardiovascular Events | | | |
| Gastro-intestinal Events | | | |
| Genito-urinary Events | | | |
| Cancer | | | |
| Hospitalization | | | |

<sup>\*</sup>per 10,000 WY of exposure

#### Additional categories / subcategories may be added for SAEs

Table C11-2 First time users only (format see Table C11-1)

Table C11-3 Repeat/Consecutive users only (format see Table C11-1)

Table **C11-**4 BMI <20 (format see Table **C11-**1)

Table **C11-**5 BMI >=20 - <30 (format see Table **C11-**1)

Table **C11-**6 BMI >=30 (format see Table **C11-**1)

Table **C11-**7 Age <30 (format see Table **C11-**1)

Table **C11-**8 Age >=30 (format see Table **C11-**1)

Table **C11**-9ff by History of respective disease (format see Table **C11**-1)

#### Table C12- Effect of Prognostic Factors on Outcomes of Interest (Date of analysis: ...)

The quantitative impact (relative risks) of potential prognostic factors on the outcomes of interest (e.g., implant palpability reported by physician, more frequent SAEs) presented in Tables C1 – C11 will be analyzed using multivariate regression models if there are at least 5 events per cell. The choice of the regression model will depend on the data: logistic regression will be used for data where the outcome is a proportion, Cox for data where the outcome is a rate.

Predefined covariates are .age (< 30 vs. ≥30yrs), BMI (<30 vs. ≥30), user status (first time users vs. repeat users), experience of healthcare professional with Implanon insertions in the past year (<10/y vs. >=10/y) and Nexplanon insertions in total (<5 NXPL vs. >=5 NXPL). Additional prognostic factors and classification categories might be added on request of regulatory authorities or the Safety Monitoring and Advisory Board. The relative risks will be presented in the following format.

| Outcome of interest | Prognostic Factor | RR | 95% CI |
|-----------------------|---------------------------|----|--------|
| Outcome of interest 1 | | | |
| | Age | | |
| | BMI | | |
| | User status | | |
| | Experience with Implanon | | |
| | Experience with Nexplanon | | |
| Outcome of interest 2 | | | |
| | Age | | |
| | BMI | | |
| | User status | | |
| | Experience with Implanon | | |
| | Experience with Nexplanon | | |
| Outcome of interest | | | |